CLINICAL TRIAL: NCT02719756
Title: Randomized, Open Prospective Study of the Effect of SGLT-2 Inhibitor Dapagliflozin on Glycemic Variability in Patients With Diabetes Mellitus Type 2
Brief Title: Effect of SGLT-2 Inhibitor Dapagliflozin on Glycemic Variability in Patients With Diabetes Mellitus Type 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Research Clinical Centre of the Russian Railways, JSC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ESR-15-11023
Record Dates: First submitted 2016-03-09; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus; Hypoglycemic Episodes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin & Dapagliflozin (Experimental): Metformin stable dose tablets and Dapagliflozin 10 mg tablets by mouths, once daily in morning for 3 months
  Interventions: Drug: Metformin; Drug: Dapagliflozin
- Metformin up-titration (Active Comparator): Metformin tablets up-titration by mouths, for 3 months
  Interventions: Drug: Metformin; Drug: Metformin up-titration

INTERVENTIONS:
Drug: Metformin — Metformin tablets 1000 mg
  Other Names: GLUCOPHAGE
Drug: Dapagliflozin — Dapagliflozin 10 mg tablets
  Other Names: FORXIGA; FARXIGA
  Arms: Metformin & Dapagliflozin
Drug: Metformin up-titration
  Arms: Metformin up-titration

SUMMARY:
This study will test the hypothesis that early use of combination therapy with dapagliflozin and metformin will provide good glycemic control with low glycemic variability and without hypoglycemic episodes, and will be better tolerated than up-titration of metformin monotherapy. The study will also correlate these benefits with glycated hemoglobin.

DETAILED DESCRIPTION:
Type 2 diabetes is a progressive, chronic metabolic disease characterized by hyperglycemia. Despite therapeutic advances, the incidence and prevalence of diabetes continue to surge. Worldwide, the number of individuals with diabetes is projected to rise from 366 million in 2011 to 552 million by 2030, which is the equivalent of approximately three new cases being diagnosed every 10 seconds. Type 2 diabetes doubles the risk of cardiovascular disease, and macrovascular complications (myocardial infarction and stroke) are a common cause of death in patients with type 2 diabetes. The U.K. Prospective Diabetes Study showed that every 1% absolute decline in mean A1C was associated with a 37% reduction in the risk of microvascular complications and a 21% reduction in the risk of any diabetes-related complication or death. Diabetes also exacts a tremendous economic burden. Meeting treatment goals is elusive for many people with diabetes. Data from the National Health and Nutrition Examination Survey from 2003 to 2006 showed that only 57.1% of adults with diagnosed diabetes achieved an A1C < 7%, 45.5% had a blood pressure level < 130/80 mmHg, and 46.5% had an LDL cholesterol level < 100 mg/dl. Only 12.2% of people with diabetes reached all three goals. Treatment of Type 2 diabetes is not limited to just glycaemic control. Rather, the proper management of hyperglycaemia, weight, blood pressure, and lipids can have benefits in terms of slowing the progression of Type 2 diabetes, decreasing the risk of CV disease, and improving overall health.Current antihyperglycaemic treatments are predominantly insulin-dependent. These treatments can effectively manage HbA1c, and treatment may be influenced by the patient's comorbidities and any potential treatment-related adverse events. However, as Type 2 diabetes progresses, regimens need to be modified to compensate for declining beta-cell function and decreasing insulin sensitivity. On this basis,the EASD/ADA guidelines suggest following a treatment pathway that has well validated therapies at it's core.Of the many comorbid conditions described, excess weight is especially important, not only because of the increased disease risk, but also for the management of blood pressure and lipids. Consequently, AACE/ACE algorithms give priority to those regimens that have the added benefit of minimising hypoglycaemic events and weight gain.In addition, while antidiabetic treatments tend to focus on insulin-dependent mechanisms in organs such as the liver and pancreas, it should not be forgotten that the kidneys also have a role in maintaining glucose homeostasis There are multiple barriers to achieving optimal glycemic control. Current medications for type 2 diabetes have potential adverse effects; for example, can cause hypoglycemia and weight gain. Hypoglycaemia is a limiting factor in the glycaemic management of patients with advanced Type 2 diabetes.Most often hypoglycaemia is associated with mild to severe neurologic symptoms, and in some cases it can result in death. Additionally, the risk of cardiac ischaemia is increased in Type 2 diabetes patients with symptomatic or asymptomatic hypoglycaemia compared with patients with hyperglycaemia or stable normoglycaemia. The risk of hypoglycaemia increases with advancing age, polypharmacy, later stages of disease, and intensive antihyperglycaemic treatment with certain drugs, such as sulphonylureas. Intensive treatment (target HbA1c<7.0%) results in a greater number of patients experiencing severe hypoglycaemic events (3-21%) compared with conventional treatment (target HbA1c ≥7.0%; 2-10%), although intensive therapy may have a greater beneficial effect in terms of a decreased risk of microvascular disease. As a result, hypoglycaemia is one of several factors, including weight gain and increases in CV disease-related and overall mortality, that may limit the microvascular benefits of intensive therapy. Thus, the search continues for novel therapeutic agents that can help patients avoid these limiting side effects while providing glycemic control.

ELIGIBILITY:
Inclusion criteria

The subject population that will be observed in the study, must fulfil all of the following criteria:

1. Signed informed consent.
2. Written informed consent by women of childbearing age to interception during study participation period, with determination of level of chorionic gonadotropic hormone by the pregnancy test, prior to study enrollment.
3. Age >=18 - 74 years.
4. eGFR >=60 mL/min/1.73 m2 by MDRD formula.
5. BMI <40 kg / m2
6. C-peptide >= 1 ng/ml
7. HbA1c 7 - 9% both included
8. Stabile 1000 mg dose of Metformin daily for at least 8 weeks prior to enrollment

Exclusion criteria

1. The presence of absolute contraindications to therapy by SGLT-2 inhibitor Dapagliflozin:

   1.1. Individual idiosyncrasy of any drug component.

   1.2. Type 1 diabetes.

   1.3. Diabetic ketoacidosis.

   1.4. Renal disease, medium to severe (eGFR <60 ml/min /1.73m2 by MDRD formula) or end-stage renal failure.

   1.5.Hereditary lactose intolerance, lactase deficiency, and glucose and galactose intolerance.

   1.6. Pregnancy and breast-feeding.

   1.7. Children under 18 years of age.

   1.8. Patients receiving loop diuretics or with reduced volume of blood circulation, such as a result of acute diseases (e.g. gastrointestinal problems).

   1.9. Elderly patients aged 75 years and older.
2. A history of moderate or severe congestive heart failure (New York Heart Association [NYHA] Class III or IV) within 3 months prior to the screening visit
3. Increased liver transaminases ALT and/or AST more than 3 times higher than normal.
4. Any condition that in the opinion of the PI confound the evaluation and interpretation of efficacy and or safety data. Significant medical or psychological condition that, in the opinion of the Investigator, would compromise the patient's safety or successful participation in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Dynamics (delta from the baseline) of blood glucose variability - integral index of glycemia (LBGI-HBGI) after 3 months of therapy | 3 months

SECONDARY OUTCOMES:
Dynamics (delta from the baseline or % decrease of blood glucose level) of blood glucose variability (ADRR) after 3 months of therapy | 3 months
Dynamics of MAGE after 3 months of therapy | 3 months
Dynamic of glycaemia parameters: % of normoglycemia time after 3 months of therapy | 3 months
Dynamic of glycaemia parameters: % of hyperglycemia time after 3 months of therapy | 3 months
Dynamic of glycaemia parameters: % of hypoglycemia time after 3 months of therapy | 3 months
Dynamics of HbA1c (%) from baseline after 3 months of therapy | 3 months
Percentage of diabetes mellitus patients achieved individual target HbA1c | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ametov, prof., MD, Principal Investigator — Research Clinical Center of the Russian Railways, JSC
Locations (1):
- Research Clinical Centre of the Russian Railways, JSC, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No